CLINICAL TRIAL: NCT00609609
Title: A Randomized Phase II Study for the Evaluation of Extracorporeal Photopheresis (ECP) in Combination With Corticosteroids for the Initial Treatment of Acute Graft-Versus-Host Disease (GVHD)
Brief Title: Photopheresis for the Treatment of Acute Graft Versus Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-1022; NCI-2012-01751 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-01-23; First posted 2008-02-07 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Graft Versus Host Disease
Keywords: Allogeneic stem cell grafts; Allogeneic bone marrow graft; Blood and Marrow Transplantation; Stem cell graft; Graft Versus Host Disease; GVHD; Extracorporeal Photopheresis; ECP; Photopheresis; Methylprednisolone; Medrol; Depo-Medrol; Solu-Medrol
MeSH Terms: conditions — Graft vs Host Disease | interventions — Photopheresis; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corticosteroids (Experimental): Methylprednisolone at a dose of 2 mg/kg/day with a taper to no less than 1 mg/kg/day by day 14, and no less than 0.4 mg/kg/day by day 28.
  Interventions: Drug: Methylprednisolone
- ECP + Corticosteroids (Experimental): Extracorporeal Photopheresis (ECP) 8-9 treatments weekly for days 1-14, 6 treatments weekly from days 15-28, and after that 2 treatments weekly until day 60 + Methylprednisolone at a dose of 2 mg/kg/day with a taper to no less than 1 mg/kg/day by day 14, and no less than 0.4 mg/kg/day by day 28.
  Interventions: Procedure: Photopheresis; Drug: Methylprednisolone

INTERVENTIONS:
Procedure: Photopheresis — 8-9 photopheresis treatments weekly for days 1-14, 6 treatments weekly from days 15-28, and after that 2 treatments weekly until day 60. After day 60, your doctor will decide whether ECP is worth continuing, and the frequency of treatments.
  Other Names: Extracorporeal Photopheresis; ECP
  Arms: ECP + Corticosteroids
Drug: Methylprednisolone — 2 mg/kg daily with a taper to no less than 1 mg/kg/day by day 14, followed by a tapering schedule according to the suggested guidelines.
  Other Names: Medrol; Depo-Medrol; Solu-Medrol

SUMMARY:
The goal of this clinical research study is to find out whether adding extracorporeal photopheresis (ECP) to standard therapy for acute GVHD with corticosteroids improves response to treatment, length of treatment, and survival.

DETAILED DESCRIPTION:
ECP uses ultraviolet A radiation to treat lymphocytes. Although the exact reason why ECP may be beneficial is not completely understood, researchers believe that the lymphocytes treated this way are less likely to continue causing GVHD.

In this study, researchers want to evaluate whether adding another treatment to standard therapy with corticosteroids, in this case ECP, will improve the response to therapy, duration of therapy, and survival. After the diagnosis of acute GVHD, you will be randomly selected (at the toss of a coin) to be in one of 2 treatment groups. One group will receive treatment with corticosteroids (like methylprednisolone or prednisone) alone, and the other will receive ECP treatments in addition to the corticosteroids. ECP treatments are explained below.

In order to have ECP, you will need a special central venous catheter similar to the one you have now. A central venous catheter is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your physician will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure.

Blood is drawn by a machine called "photopheresis machine". This blood goes into a bowl inside the machine, where it is spun and separated into white cells (called buffy coat), red cells, and platelets. The red cells and platelets are promptly returned to you, while the white cells in the buffy coat undergo the process of ECP. The buffy coat will come out of the bowl and will be mixed with a substance called methoxsalen, that will make lymphocytes more sensitive to the effects of light. After mixing with methoxsalen, the buffy coat goes in to chamber where it is exposed to ultraviolet A radiation, and from there back to you. This process is done gradually, in cycles, and takes about 3 hours.

You will have up to 4 of these treatments weekly for the first 14 days of therapy, then 3 treatments weekly from Day 15-28, and after that 2 treatments weekly until Day 60, which is the end of the study. After Day 60, your doctor will decide whether ECP is worth continuing, and also the frequency of treatments. It is not necessary to be in the study to continue to receive ECP treatments. If you respond to the treatment, your corticosteroids will be reduced slowly to prevent the GVHD from coming back.

The length of corticosteroid therapy will depend on how GVHD responds to the treatment. You will follow a corticosteroid therapy tapering schedule according to the suggested guidelines. You will continue to receive tacrolimus or cyclosporine, whichever you have been using as GVHD prevention, throughout the study independent of what treatment group you are assigned.

While you are getting treatment in this study, every week you will have a physical exam and blood (about 1 tablespoon) will be drawn for routine tests. If your doctor thinks it is necessary, blood may be drawn more often.

You will be considered off-study after 6 months of treatment completion. You will be taken off study if you are unable to comply with study requirements, you refuse to continue participation in the study, or intolerable side effects occur.

This is an investigational study. ECP has been approved by the FDA for the treatment of a certain type of lymphomas of the skin and is commercially available. Its use in patients with GVHD is considered to be investigational. Up to 95 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be recipients of allogeneic bone marrow or stem cell grafts.
2. Patient must weigh above 40 kg
3. Patients must have new onset, clinical grade II-III acute or late-acute GVHD of the GI tract or liver, or the skin that developed post transplantation. The diagnosis of GVHD must be pathologically confirmed in at least one organ or highly suspected clinically. Pathological confirmation may occur after registration and after the start of therapy. Definition of Late Acute GVHD vs Acute GVHD: The diagnosis of Late Acute GVHD includes clinical features that are identical to Acute GVHD, however, Late Acute GVHD is diagnosed on or after day 100 post transplantation.
4. Continued from #3: These manifestations include a maculopapular rash, abnormal liver studies (cholestatic jaundice) and/or nausea/vomiting / diarrhea. Patients must not have any concurrent classical features of chronic GVHD in addition to the above manifestations. Features of chronic GVHD include dry eyes and mouth, contractures, and/ or sclerodermal, lichenoid skin changes.
5. In the clinical judgment of the PI, patients must be able to sustain a platelet count and a hematocrit >/= 20,000/mL and >/= 27% respectively, with or without transfusions.
6. The absolute white blood cell count (WBC) must be >1500/mL
7. Patient must be willing to comply with all study procedures.
8. All patients with childbearing potential, including males and females, must commit to using adequate contraceptive precautions throughout their participation in the study and for 3 months following the last ECP treatment.

Exclusion Criteria:

1. Patients developing chronic GVHD following immune modulation with immunosuppression withdrawal or donor lymphocyte infusion (DLI).
2. Any clinical Manifestation consistent with de novo chronic GVHD or overlapped syndrome of acute and chronic GVHD.
3. Patients who are unable to tolerate the volume shifts associated with ECP treatment due to the presence of any of the following conditions: uncompensated congestive heart failure, pulmonary edema, severe asthma or chronic obstructive pulmonary disease, hepatorenal syndrome.
4. Active bleeding
5. International normalized ration (INR) >2
6. Patients cannot have received methylprednisolone > 2mg/kg/day for more than 72 hours prior to registration.
7. Patients cannot have received any other immunosuppression for treatment of GVHD but calcineurin inhibitors and corticosteroids. Patients are allowed to have had any GVHD prophylaxis with the exception of ECP
8. Patients with known hypersensitivity or allergy to psoralen
9. Patients with known hypersensitivity or allergy to both citrate and heparin
10. Patients with co-existing photosensitive disease (e.g. porphyria, systemic lupus erythematosus, albinism) or coagulation disorders.
11. Uncontrolled, persistent hypertriglyceridemia, with levels > 800 mg%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amin Alousi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 23, 2008 to November 19, 2014. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Corticosteroids | ECP + Corticosteroids
Started | 30 | 51
Completed | 24 | 49
Not Completed | 6 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Progression | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corticosteroids | ECP + Corticosteroids | Total
Number analyzed (Participants) | 30 | 51 | 81
Age, Continuous [Median (Full Range); unit: years] | 53 [24 to 70] | 54 [17 to 75] | 54 [17 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 20 | 31
  Male | 19 | 31 | 50
Region of Enrollment [Number; unit: participants]
  United States | 30 | 51 | 81
Ablative Conditioned [Count of Participants; unit: Participants] | 23 | 33 | 56
GVHD Prophylaxis [Count of Participants; unit: Participants]
  Tacrolimus/MTX | 28 | 44 | 72
  Tacrolimus/Mycophenolate | 0 | 5 | 5
  Other | 2 | 2 | 4
Donor Relation [Count of Participants; unit: Participants]
  Related | 12 | 18 | 30
  Unrelated | 18 | 33 | 51
Donor Match [Count of Participants; unit: Participants]
  Matched | 24 | 41 | 65
  Mismatched/Haploidentical | 6 | 10 | 16
Graft Source [Count of Participants; unit: Participants]
  Peripheral Blood | 25 | 36 | 61
  Bone Marrow | 5 | 10 | 15
  Umbilical Cord | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Day 56 Treatment Success
Description: Definition of Treatment Failure: No Response according to the following: A) Skin: 1) No change in GVHD stage by day 14; 2) Gut: No change in GVHD stage by Day 7; 3) Liver: No change in GVHD stage by Day 21. B) Progressive Disease (PD): 1) Skin/Gut: Increase in Stage by 72 hours from the start of therapy; 2) Liver: Increase in Stage by Day 14; 3) Initiation of 2nd line treatment at any time for acute GVHD: 4) Any new organ involvement by acute GVHD. C) Inability to Taper: 1) Patient still on >1 mg/kg/d of methylprednisolone equivalent at 1 month. 2) Patient still on > 0.5 mg/kg/d of methylprednisolone equivalent at 2 months; 3) Death from GVHD. Definition of Treatment Success: Participants not defined above in Treatment Failure definition. Baseline biopsy with Acute GVHD assessed weekly until last ECP procedure (anticipated Day 63). At 6 months follow up with a phone call for survival and GVHD status.
Time Frame: Day 1 to Day 63 (approximately 9 weeks), Acute GVHD scored weekly.
Measure: Number; unit: percentage of participants
Arm/Group | Corticosteroids | ECP + Corticosteroids
Number analyzed (Participants) | 30 | 51
percentage of participants
  Skin-only | 57 | 72
  Visceral Involvement | 43 | 47
  Total | 53 | 65

2. Post Hoc Outcome: Percentage of Participants Alive, In Remission & Without GVHD Progression Day 28 & Day 56
Description: Percentage meeting steroid milestone who were alive, in remission and did not have GVHD progression before Day 28 or Day 56.
Time Frame: Up to day 56
Measure: Number; unit: percentage of participants
Arm/Group | Corticosteroids | ECP + Corticosteroids
Number analyzed (Participants) | 30 | 51
percentage of participants
  Day 28 Steroid dose </= 0.25mg/kg | 10 | 23.5
  Day 56 steroid dose < 0.1mg/kg | 30 | 43

3. Post Hoc Outcome: Non-relapse Mortality (NRM) at 6 Months
Description: Percentage of participants at 6 months whose deaths were without relapse/recurrence.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Corticosteroids | ECP + Corticosteroids
Number analyzed (Participants) | 30 | 51
percentage of participants | 19.6 [8.6 to 30.6] | 20.0 [5.4 to 34.6]

ADVERSE EVENTS:
Time Frame: Adverse events collected through weekly treatments for up to 60 days.
Arm/Group | Corticosteroids | ECP + Corticosteroids
Serious Adverse Events (participants affected / at risk) | 4/30 | 4/51
Other Adverse Events (participants affected / at risk) | 30/30 | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corticosteroids (N=30) | ECP + Corticosteroids (N=51)
Graft versus Host Disease (GVHD) (General disorders) | 0 (0) | 1 (1)
Refractory GVHD (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Liver Failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Multi-system organ failure (General disorders) | 0 (0) | 1 (1)
GI GVHD (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corticosteroids (N=30) | ECP + Corticosteroids (N=51)
acute kidney injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
acute renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Altered mental status (Psychiatric disorders) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
aspergillus pneumonia infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
bilateral pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BK virus infection (Infections and infestations) | 4 (4) | 6 (6)
bladder spasms (Renal and urinary disorders) | 0 (0) | 1 (1)
candida albicansfungus infection (Infections and infestations) | 0 (0) | 1 (1)
candida glabrata pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
catheter related mycobateremia (Surgical and medical procedures) | 0 (0) | 1 (1)
Cytomegalovirus (CMV) infection (Infections and infestations) | 5 (5) | 11 (11)
Central Nervous System (CNS) ischemia (Nervous system disorders) | 0 (0) | 1 (1)
cystitis (Renal and urinary disorders) | 0 (0) | 3 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
delayed infusion reactions (Surgical and medical procedures) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
dysuria (Renal and urinary disorders) | 0 (0) | 2 (2)
e. coli urinary tract infection (UTI) (Infections and infestations) | 1 (1) | 1 (1)
edema (General disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (elevated ALT) (Investigations) | 0 (0) | 4 (4)
Aspartate transaminase increased (AST) (Investigations) | 0 (0) | 1 (1)
elevated bilirubin (Investigations) | 0 (0) | 2 (2)
elevated creatinine (Investigations) | 0 (0) | 2 (2)
enterococcus infection (Infections and infestations) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
flu-like symptoms (General disorders) | 1 (1) | 0 (0)
GI bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI Graft versus Host Disease (GVHD) (Gastrointestinal disorders) | 0 (0) | 2 (2)
gram positive cocci infection (Infections and infestations) | 1 (1) | 0 (0)
ground glass opacity bilateral lungs (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
hemorrage (General disorders) | 0 (0) | 1 (1)
herpes infection (Infections and infestations) | 0 (0) | 2 (2)
HHV6 infection (Infections and infestations) | 1 (1) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
increase creatinine (Investigations) | 0 (0) | 1 (1)
infection (Infections and infestations) | 2 (2) | 1 (1)
influenza infection (Infections and infestations) | 1 (1) | 0 (0)
Liver Graft versus Host Disease (GVHD) (Hepatobiliary disorders) | 0 (0) | 1 (1)
muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
norovirus infection (Infections and infestations) | 0 (0) | 1 (1)
ocular gvhd (Eye disorders) | 1 (1) | 1 (1)
parafluenza pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Parvovirus (Infections and infestations) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
peritoneal fluid infection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
polymicrobial infection (Infections and infestations) | 0 (0) | 1 (1)
pseudomonas aeruginosa bacteremia (Infections and infestations) | 0 (0) | 3 (3)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Renal dysfunction (Renal and urinary disorders) | 1 (1) | 1 (1)
Respiratory effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RSV pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
sepsis (Infections and infestations) | 0 (0) | 1 (1)
skin rash (Skin and subcutaneous tissue disorders) | 3 (3) | 9 (9)
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
staphylococcus infection (Infections and infestations) | 2 (2) | 4 (4)
staphylococcus lower respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
thrombosis (Vascular disorders) | 1 (1) | 4 (4)
Thrombotic microangiopathy (Vascular disorders) | 1 (1) | 0 (0)
toe pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
urine staphylococcus infection (Renal and urinary disorders) | 2 (2) | 3 (3)
Vancomycin resistent enterococci infection (Infections and infestations) | 0 (0) | 2 (2)
Vascular obstruction (Vascular disorders) | 0 (0) | 1 (1)
Hepatic veno-occlusive disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
viral encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes